CLINICAL TRIAL: NCT04009486
Title: Impact of Whole Body Vibration on Sleep Symptoms and the Brain in Obstructive Sleep Apnea
Brief Title: Whole Body Vibration and the Brain in OSA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not approved for funding
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-006112
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obstructive Sleep Apnea (Experimental): Subjects will undergo 6 weeks of whole body vibration.
  Interventions: Device: Whole Body Vibration

INTERVENTIONS:
Device: Whole Body Vibration — Subjects will undergo whole body vibration (standing on a "power plate" device 3 times a week, for 30 minute sessions, for 6 weeks)

SUMMARY:
Participants will have an overnight polysomnography (recording apnea-hypopnea index), MRI (brain structure), and a sleep symptoms questionnaire for baseline data. Participants will then undergo 6 weeks of whole body vibration (using the whole body vibration device), 3 times a week for 30 minutes sessions. After 6 weeks, participants will have complete another polysomnography, MRI and sleep questionnaire.

DETAILED DESCRIPTION:
OSA subjects will be recruited from the UCLA Sleep Disorders Center via recruitment flyers. When prospective subjects contact the study coordinator, the study will be explained in greater detail, and inclusion and exclusion criteria reviewed. If the person agrees to participate, appointments for data collection will be made and copies of the informed consent will be mailed for their review for at least 3 days before the study. Then the Project Coordinator or one of the PI's will contact the prospective subject, answer any questions about the study, and obtain signed, informed consent. Baseline measures (PSQI, BDI-II, height, weight, vital signs [temperature, heart rate, blood pressure]) will be obtained. At 6 weeks, baseline measures will be repeated and an overnight polysomnography study will be performed at the subject's home. All subjects will be given the WBV device at the end of the study. Delivery of the WBV device to each subject's home will be arranged and the WBV device and pedometer set up by the research team. Training in the use of the WBV device will be provided inperson and via written instructions. Phone and e-mail support for the WBV device or any study questions will be available for all study participants. Subjects will use the device at least 3 times/week, for 30 minutes per session, for 6 weeks. In addition to the pedometer, a wall calendar will be provided on which subjects will mark the days that they use the WBV device. Project Coordinator will visit subjects weekly, and as needed, to record pedometer readings, check wall calendar for WBV device use, and to answer any subjects' questions or concerns. Brain MRI scans will be performed at baseline and after 6 weeks. An MRI-compatible pulse oximeter, and an air-filled pressure transducer will be connected to the subject to monitor heart rate, O2 saturation, and thoracic wall movement, and then the subject will be positioned in the scanner for data collection.

ELIGIBILITY:
Inclusion Criteria:

* AHI ≥15
* new diagnosis of moderate to severe OSA (via overnight polysomnography)
* and able to lay flat (requirement for brain MRI)
* must have space and electrical power access for WBV device at their home

Exclusion Criteria:

* other forms of sleep-disordered breathing (such as central sleep apnea, restless legs syndrome, mixed sleep apnea)
* currently using (or will start using during 6-week study period) CPAP or BiPAP or oral appliance for OSA treatment
* recent (<6 months) myocardial infarction
* current pregnancy (if subject is female)
* history of stroke
* diagnosed psychiatric disease (schizophrenia, manic-depressive)
* airway or chest deformities that would interfere with breathing
* mechanical ventilatory support
* renal failure (requiring dialysis)

For brain MRI

* claustrophobia
* metallic-based tattoos
* metallic implants or devices (such as implantable cardioverter-defibrillator, pacemaker, embolic coils, aneurysm clips) or any other material that could be hazardous in MRI scanner
* body weight >300 lbs (restrictions of MRI scanner table)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | after 6 weeks of whole body vibration use
  average number of times per hour during the sleep study/overnight polysomnography that the subject's arterial blood oxygen saturation drops by over 10% from waking baseline

SECONDARY OUTCOMES:
Sleep Symptoms | after 6 weeks of whole body vibration use
  symptoms associated with sleep disturbances within the previous month, as recorded by the Pittsburgh Sleep Quality Index Questionnaire (measures sleep symptoms, such as fatigue, sleep quality, sleep duration, etc.The PSQI is a 19-item self-report questionnaire which queries the subject regarding sleep symptoms for the month before the instrument's administration. Each question is rated on a 0-3-point scale, with a total score range of 0-21. Higher scores indicate worse sleep symptoms. A global sum of > 5 indicates a "poor" sleeper. The PSQI has good validity when compared with overnight polysomnography measures and acceptable reliability (Cronbach's alpha > 0.7; test-retest reliability 0.72-0.86)
Brain Structure | after 6 weeks of whole body vibration use
  high resolution T1 or T2 (diffusion tensor imaging) examination of brain structure changes (baseline and after 6 weeks)